CLINICAL TRIAL: NCT01654887
Title: Comparative Effectiveness of Lung Ultrasound vs. Chest X-ray for the Diagnosis of Pneumonia in the Emergency Department
Brief Title: A Randomized Controlled Trial of Lung Ultrasound Compared to Chest X-ray for Diagnosing Pneumonia in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 12-0428; HSM# 12-00153
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Pneumonia
Keywords: Comparative Effectiveness; Lung Ultrasound versus Chest X-ray; Pneumonia; Emergency Department
MeSH Terms: conditions — Pneumonia; Emergencies | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lung Ultrasound (Experimental): LUS first with the option of obtaining CXR second
  Interventions: Other: Lung Ultrasound
- Chest X-Ray (Active Comparator): CXR first followed by LUS second
  Interventions: Radiation: Chest X-Ray

INTERVENTIONS:
Other: Lung Ultrasound — Six anatomic areas, delineated by the anterior, posterior, and mid- axillary lines will be systematically examined bilaterally, as per the modified Bedside Lung Ultrasound in Emergency (BLUE) protocol (Lichtenstein 2008). Ultrasound images will be obtained in longitudinal and transverse orientation, and recorded.
  Other Names: LUS
  Arms: Lung Ultrasound
Radiation: Chest X-Ray — Posterior-Anterior and lateral views of the chest via chest radiography followed by a lung ultrasound which is comprised of six anatomic areas, delineated by the anterior, posterior, and mid- axillary lines will be systematically examined bilaterally, as per the modified Bedside Lung Ultrasound in Emergency (BLUE) protocol (Lichtenstein 2008). Ultrasound images will be obtained in longitudinal and transverse orientation, and recorded.
  Other Names: CXR
  Arms: Chest X-Ray

SUMMARY:
The primary objective of this study is to determine if lung ultrasound (LUS) can replace chest x-ray (CXR) when evaluating patients with possible pneumonia. Specifically, we are looking for an overall reduction of CXR when LUS is used first. Our null hypothesis is that LUS cannot replace CXR for diagnosing pneumonia. Our alternate hypothesis is that LUS can replace CXR for diagnosing pneumonia. Our secondary objectives include: (1) a comparison of unscheduled healthcare visits after the index Emergency Department (ED) visit between those subjects who undergo CXR first and those who undergo LUS first, (2) an evaluation of the rate of antibiotic use between the two groups, (3) a comparison of the admission rates, and (4) a comparison of the length of stay in the Emergency Department between the two groups.

DETAILED DESCRIPTION:
Background - Ultrasound is now widely accepted as a diagnostic tool for use in the emergency department, as supported by the American College of Emergency Physicians position statement in 2001 (revised in 2008). Evidence-based guidelines for point-of-care lung ultrasound have recently been published (Volpicelli et al 2012). Lichtenstein et al (2004) performed bedside LUS on 117 critically ill patients to evaluate for alveolar consolidation and compared these findings with CT, the gold standard. Sensitivity of ultrasound was 90% and specificity 98%, indicating that US is a feasible imaging modality for the lungs. Copetti et al (2008) compared the diagnostic accuracy of LUS and CXR in children with suspected pneumonia. 79 children underwent LUS and CXR. Lung ultrasound was positive for the diagnosis of pneumonia in 60 patients, whereas CXR was positive in 53. Copetti concluded that LUS is as reliable as CXR in diagnosing pneumonia plus it has the added benefit of no radiation exposure for patients. Shah et al (2009) found LUS to be superior to CXR in detecting pneumonia. 200 patients with suspected pneumonia were enrolled and underwent LUS and CXR. LUS detected 49 pneumonias whereas CXR detected 36. The 13 cases of radiographically occult pneumonia that were identified by LUS were all less than 1 centimeter in diameter, suggesting that LUS is superior in identifying early and/or small pulmonary consolidations. This particular study found that LUS was able to detect pneumonia with a Sensitivity of 86% and a Specificity of 97%. Additionally, Tsung et all (2009) found that it is feasible to use ultrasound to distinguish viral from bacterial pneumonia, thus indicating another striking advantage to LUS. From these studies, it is clear that lung ultrasound plays a role in the diagnosis of pulmonary pathology and moreover it is possible that LUS may replace CXR as the imaging modality of choice. This study is designed as a comparative effectiveness randomized controlled trial between ultrasound and chest x-ray for diagnosing pneumonia. The study cited above performed by Shah et al 2009 forms the basis of our pilot data in planning this randomized controlled trial. In Dr. Shah's study, there were no missed pneumonias and no over or under treatment of pneumonia when pneumonia was diagnosed on lung ultrasound.

Study Design - Currently CXR is the standard of care for the detection of pneumonia, however, there is published evidence that demonstrates LUS is as reliable as CXR and even surpasses CXR in detecting small and/or early pneumonias as well differentiating viral from bacterial processes as cited above (Lichtenstein et al 2004; Copetti et al 2008; Shah et al 2009; Tsung et al 2012).

The motivation for conducting this study is that we have possibly identified an imaging modality that is better than our current standard of care. It is our primary aim to compare the two imaging modalities to clinical outcomes to see if subjects in the investigational arm have better outcomes than those in the control arm who receive the standard of care.

The attending physician or fellow caring for the patient will determine if the patient is eligible. If the ED provider clearly identifies a pneumonia on the ultrasound then the patient will be diagnosed and treated for pneumonia without being subjected to the unnecessary radiation of a CXR. However, if the provider does not clearly identify a pneumonia on ultrasound or if the LUS fails to detect a pneumonia and the clinical suspicion remains high, then the provider has the option to proceed to the CXR to assist in the diagnosis of pneumonia. Alternatively, all subjects randomized to the control arm will under a CXR first followed by a LUS, because LUS can often provide additional information that CXR does not as noted above (e.g. the ability to differentiate between viral and pneumonia infections).

ELIGIBILITY:
Inclusion Criteria:

* All patients who present to the ED with respiratory symptoms suspicious for pneumonia
* In whom the treating physician believes would benefit from diagnostic imaging

Exclusion Criteria:

* Patients who arrive at the ED with a previously performed CXR
* Unstable patients with life-threatening injuries who require ongoing resuscitation

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 191 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Tsung, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Emergency Ultrasound Guidelines. Policy Statement by the American College of Emergency Physicians (revised in October 2008)
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Lichtenstein DA, Lascols N, Meziere G, Gepner A. Ultrasound diagnosis of alveolar consolidation in the critically ill. Intensive Care Med. 2004 Feb;30(2):276-281. doi: 10.1007/s00134-003-2075-6. Epub 2004 Jan 13. PMID 14722643
- [Background] Copetti R, Cattarossi L. Ultrasound diagnosis of pneumonia in children. Radiol Med. 2008 Mar;113(2):190-8. doi: 10.1007/s11547-008-0247-8. Epub 2008 Apr 2. English, Italian. PMID 18386121
- [Background] Shah et al. "The Feasibility of Diagnosing Pediatric Pneumonia Using Point-of-Care Ultrasound." Pediatric Emergency Care. American Academy of Pediatrics, Section on Emergency Medicine, Scientific Abstract Presentations, AAP National Conference and Exhibition, October 16, 2009 Y Washington, DC. Ped Emerg Care. Volume 25(10), October 2009, pp 704-712.
- [Background] Tsung JW, Kessler DO, Shah VP. Prospective application of clinician-performed lung ultrasonography during the 2009 H1N1 influenza A pandemic: distinguishing viral from bacterial pneumonia. Crit Ultrasound J. 2012 Jul 10;4(1):16. doi: 10.1186/2036-7902-4-16. PMID 22862998
- [Derived] Jones BP, Tay ET, Elikashvili I, Sanders JE, Paul AZ, Nelson BP, Spina LA, Tsung JW. Feasibility and Safety of Substituting Lung Ultrasonography for Chest Radiography When Diagnosing Pneumonia in Children: A Randomized Controlled Trial. Chest. 2016 Jul;150(1):131-8. doi: 10.1016/j.chest.2016.02.643. Epub 2016 Feb 26. PMID 26923626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with suspected pneumonia in an emergency department were recruited from the Pediatric Emergency Department at Mount Sinai Hospital.
Groups:
- Lung Ultrasound: Patients in the investigational arm received a LUS. If there was clinical uncertainty after ultrasound, clinicians had the option to obtain CXR.
- Chest X-Ray: Patients in the control arm underwent sequential imaging with CXR followed by LUS.
Period: Overall Study
Arm/Group | Lung Ultrasound | Chest X-Ray
Started | 103 | 88
Completed | 103 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lung Ultrasound | Chest X-Ray | Total
Number analyzed (Participants) | 103 | 88 | 191
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3 [1.6 to 6.0] | 3 [1.7 to 5.7] | 3 [1.6 to 6.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 100
  Male | 52 | 39 | 91
Tachypnea for age [Number; unit: participants] — Tachypnea - respiratory rate >60 breaths/minute in children <2 months of age, >50 breaths/minute in children 2 to 12 months of age, and >40 breaths/minute in children ≥1 year of age.
  participants
    yes | 27 | 25 | 52
    no | 76 | 63 | 139
Triage Fever >= 38 degrees celsius [Number; unit: participants]
  yes | 48 | 41 | 89
  no | 55 | 47 | 102
Cough [Number; unit: participants]
  yes | 101 | 86 | 187
  no | 2 | 2 | 4
Difficulty breathing [Number; unit: participants]
  yes | 56 | 48 | 104
  no | 47 | 40 | 87
Chest pain [Number; unit: participants]
  yes | 17 | 10 | 27
  no | 86 | 78 | 164
Abdominal pain [Number; unit: participants]
  yes | 12 | 10 | 22
  no | 91 | 78 | 169
History of fever [Number; unit: participants]
  yes | 87 | 75 | 162
  no | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants For Whom CXR Was Not Needed to Diagnose Pneumonia
Description: The percentage of Participants For Whom CXR Was Not Needed (or received only lung US) to Diagnose Pneumonia. The primary objective of this study is to determine if it is possible for lung ultrasound (LUS) to replace chest x-ray (CXR) when evaluating patients with possible pneumonia. Specifically, an overall reduction of CXR when LUS is used first. Null hypothesis is that LUS cannot replace CXR for the diagnosis of pneumonia. Alternate hypothesis is that LUS can replace CXR for pneumonia.
Time Frame: up to 5 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lung Ultrasound | Chest X-Ray
Number analyzed (Participants) | 103 | 88
percentage of participants | 38.8 [30.0 to 48.9] | 0 [0.0 to 3.6]

2. Secondary Outcome: Comparison of Unscheduled Healthcare Visits
Description: Percentage of participants who had unscheduled healthcare visits after the index Emergency Department visit between those subjects who undergo CXR first and those who undergo LUS first.
Time Frame: week 1-2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Lung Ultrasound; Chest X-Ray: Patients in the control arm underwent sequential imaging with CXR followed by LUS.
Arm/Group | Lung Ultrasound | Chest X-Ray
Number analyzed (Participants) | 103 | 88
percentage of participants | 8.7 [3.3 to 14.1] | 11.4 [4.8 to 18.0]

3. Secondary Outcome: Percentage of Participants With Antibiotic Use
Description: A chart review and follow up phone call made at 1-2 weeks to assess whether or not the subject was started on antibiotics during the index Emergency Department (ED) visit or at a later healthcare visit.
Time Frame: weeks 1-2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lung Ultrasound | Chest X-Ray
Number analyzed (Participants) | 103 | 88
percentage of participants | 37.9 [28.5 to 47.2] | 27.3 [17.9 to 36.6]

4. Secondary Outcome: Percentage of Participants Who Had Hospital Admission.
Description: Chart review and follow up phone call made at 1-2 weeks to assess whether or not the subject was admitted during the index ED visit or at a later healthcare visit.
Time Frame: weeks 1-2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lung Ultrasound | Chest X-Ray
Number analyzed (Participants) | 103 | 88
percentage of participants | 19.4 [11.8 to 27.0] | 17.0 [9.2 to 24.8]

5. Secondary Outcome: Comparison of the Length of Stay in the ED
Description: Chart review conducted to assess overall LOS in the ED.
Time Frame: up to 5 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Lung Ultrasound | Chest X-Ray
Number analyzed (Participants) | 103 | 88
minutes | 153 [120 to 252] | 180 [139 to 241]

6. Primary Outcome: Percentage of Participants Whose Pneumonia Was Missed by LUS or CXR
Time Frame: week 1-2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lung Ultrasound | Chest X-Ray
Number analyzed (Participants) | 103 | 88
percentage of participants | 0.0 [0.0 to 2.9] | 0.0 [0.0 to 3.0]

ADVERSE EVENTS:
Time Frame: Adverse event collected duration of study, up to 2 weeks.
Arm/Group | Lung Ultrasound | Chest X-Ray
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/88
Other Adverse Events (participants affected / at risk) | 0/103 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes